CLINICAL TRIAL: NCT06075446
Title: Calling All Dads! Evaluation of APAs ACT Program: Engaging Fathers to Prevent Adverse Childhood Experiences
Acronym: CAD
Status: Active, not recruiting | Type: Observational
Sponsor: Georgia State University (Other)
Responsible Party: Principal Investigator, Dennis Reidy, Associate Professor, Georgia State University
Other Study IDs: H22282; R01CE003333-01 (NIH)
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Child Abuse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Treatment: Those with an exposure.
  Interventions: Behavioral: ACT Raising Safe Kids
- Control: Those without an exposure.

INTERVENTIONS:
Behavioral: ACT Raising Safe Kids — American Psychological Association ACT Raising Safe Kids
  Other Names: ACT RSK
  Groups: Treatment

SUMMARY:
The goal of this observational study is to assess the American Psychological Association's ACT Raising Safe Kids program with male caregivers. The main question[s] it aims to answer are: • Will male caregivers in the ACT Raising Safe Kids program report lower child maltreatment, rates of interpersonal violence, and youth aggression. • Does the ACT RSK program have a positive return on investment and will children and caregivers in the ACT RSK condition have a higher quality adjusted life years. Participants will complete four surveys over time and attend the 9-week ACT Raising Safe Kids program. Researchers will compare survey responses from male caregivers taking the ACT Raising Safe Kids classes to male caregivers not taking ACT Raising Safe Kids classes to see if there are changes in anger regulation, family conflict, parent-child conflict, and relationship satisfaction.

DETAILED DESCRIPTION:
The overall goal of the proposed 3-year project is to determine the efficacy and cost-benefit of ACT Raising Safe Kids, an evidence-based child maltreatment (CM) prevention program to prevent multiple forms of violence by male caregivers and their children. The program, ACT Raising Safe Kids (ACT), was developed by the American Psychological Association and identified in the Center for Disease Control & Prevention's technical package, Preventing Child Abuse & Neglect, as a promising strategy to prevent child maltreatment. Evidence suggests the ACT program reduces coercive, harsh, and physically aggressive parenting practices; increases positive, nurturing parenting practices; and reduces children's externalizing, aggressive, bullying behavior. While suggesting the efficacy of ACT in reducing child maltreatment, existing program evaluations have been limited by the near complete absence of male caregivers in the evaluations. This is a critical gap as male caregivers are perpetrators in nearly 50% of substantiated child maltreatment cases and are more likely to engage in harsh discipline and corporal punishment that could cause injury. The true innovation of the work lies in examining the potential of ACT to additionally prevent intimate partner violence (IPV) perpetration by male caregivers and subsequent youth violence (YV) by their children. To date, no evaluation of ACT has examined the combined prevention effects on CM, IPV, and YV among men or women.

ELIGIBILITY:
Inclusion Criteria:

* Full or partial custody of a child between the ages of one and ten years. Must read English or Spanish.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Must be male.
Study Population: Adult fathers (including male caregivers and guardians) of children ages one through ten years old based in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Corporal punishment | One year post intervention.
  Measured by subscale on the Parent Child Conflict Tactics Scale.

SECONDARY OUTCOMES:
Parenting distress | One year post intervention.
  Measured by the Parenting Stress Index.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis E Rdiedy, Phd, Principal Investigator — Georgia State University School of Public Health
Locations (1):
- Georgia State University School of Public Health, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided